CLINICAL TRIAL: NCT01884987
Title: Phase II Study of Monosialotetrahexosylganglioside for Cerebral Radiation Necrosis
Brief Title: Treatment of Cerebral Radiation Necrosis With GM1, a Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Fan Ming, Professor, Fudan University
Other Study IDs: CRN2013
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Radiotherapy; Nasopharyngeal Carcinoma; Cerebral Radiation Necrosis; MRI
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — G(M1) Ganglioside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- group one will receive non-GM1 conservative therapy: Group one will receive conservative therapy such as hyperbaric therapy or corticosteroids therapy or "wait and see" policy
  Interventions: Drug: GM1

INTERVENTIONS:
Drug: GM1 — This group will be treated with GM1 80mg daily for 14 days, and then followed with GM1 40mg daily for 46 days.
  Other Names: monosialotetrahexosylganglioside

SUMMARY:
Cerebral radiation necrosis (CRN) is a well-documented late complication of radiation therapy for cancers, and may have a devastating effect on the patient's quality of life (QOL). However,CRN was once regarded as a progressive and irreversible disease, no standard therapy has been suggested for CRN. In our clinical practice, we have used monosialotetrahexosylganglioside (GM1)to treat CRN, and found that GM1 can successfully reverse CRN. So we carried out this prospective study to test the efficacy of GM1 for CRN.

ELIGIBILITY:
Inclusion Criteria:

The necrotic mass shown on MRI must be measured in two dimensions. No local or regional recurrence, no distant metastasis. Karnofsky performance status of at least 70 and were supposed to live more than 6 months.

Exclusion Criteria:

* CRN combined with local or regional relapse, or with distant metastasis. ② CRN combined with other cerebrovascular disease. ③CRN combined with the second primary malignancy. ④ CRN without neurologic symptoms or signs. ⑤ CRN combined with diabetes. ⑥CRN patients that were supposed to live less than 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have undergone definitive RT for histologically confirmed NPC years before. They were required to have at least two consecutive magnetic resonance imaging (MRI) study supporting the diagnosis of CRN with an interval of 3-4 months, with the second MRI showing progressive disease compared with the first MRI. The necrotic mass shown on MRI must be measured in two dimensions in order to define the response to treatment. Other radiologic studies were also required to support the non-existence of local or regional recurrence, distant metastasis. Patients must have undergone mental status examinations and had progressive neurologic symptoms or signs. In addition, they were required to have a Karnofsky performance status of at least 70 and were supposed to live more than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The necrotic volume showed on MRI | 6-8 months

SECONDARY OUTCOMES:
relief of the symptoms related to CRN | 6-8 months

CONTACTS AND LOCATIONS:
Overall Officials: ChaoSu Hu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Cancer Center, Fudan University, Shanghai, China